CLINICAL TRIAL: NCT00542061
Title: Clinical Effectiveness and Cost-effectiveness of a Monitoring System for Patients With COPD and Asthma With Persistent Obstruction in Primary Care; a Multicentre Randomised Nested Clinical Trial
Brief Title: Monitoring Asthma and COPD in Primary Care
Acronym: Monaco
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: PICASSO: Partners in Care Solutions for COPD (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Picasso 04-008
Record Dates: First submitted 2007-10-08; First posted 2007-10-10 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2007-10

CONDITIONS: Lung Diseases, Obstructive; Asthma
Keywords: COPD; Asthma; Lung function; Monitoring; Primary Care
MeSH Terms: conditions — Lung Diseases, Obstructive; Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Device: monitoring services
  Interventions: Device: half-yearly monitoring routine
- B (No Intervention): Control group: no monitoring procedures

INTERVENTIONS:
Device: half-yearly monitoring routine — A written expert advice for GPs on additional diagnostic, treatment, and referral of patients with asthma and COPD based on half-yearly monitoring routines (lung function assessments including extensive anamnese) supported by half-yearly visits of an AC nurse consultant to the general practices.
  Arms: A

SUMMARY:
The purpose of this study is to determine the clinical effectiveness and cost-effectiveness of a written expert advice for GPs on additional diagnostic, treatment, and referral of patients based on half-yearly monitoring routines for patients with COPD or ashtma with a persistent obstruction in primary care based on a multicentre randomised nested clinical trial

DETAILED DESCRIPTION:
In the Netherlands, the majority of patients (60-80 %) with asthma or COPD are treated in primary care, primarily by General Practitioners (GPs). In 1995 a Regional Diagnostic Centre, Etten-Leur, The Netherlands (also called SHL: Stichting Huisartsen Laboratorium) started a lung function monitoring service for patients with asthma and COPD of GPs in the region. The GP receives recommendations on treatment, additional diagnostics and referrals of the patient based on extensive anamnesis (i.e. dyspnoea, symptoms, smoking stage), measurement of lung function, and BMI. Moreover,the general practitioners are supported by an Asthma/COPD nurse that visit the general practice half-yearly.

Main research question of this study: Is a written expert advice for GPs on additional diagnostic, treatment, and referral of patients based on half-yearly monitoring of patients with COPD or asthma with a persistent airway obstruction with support of an AC nurse consultant related to less impaired health related quality of life (HRQoL), less symptoms and better lung function of the patients compared to usual care?

A multi-centre, single blinded (patient, lung function assistant, advisor, and research team are blinded), parallel group study is carried out to compare the monitoring intervention with usual care during 24 months. General practices were allocated by a minimisation procedure and all participating patients of a general practice were allocated to the same treatment group (nested design).

ELIGIBILITY:
Inclusion Criteria:

* The patient is categorised as asthmatic disease with persistent airway obstruction or COPD in the monitoring system SHL confirmed by the most recent lung function assessment (FEV1/FVC < 70% after BD and FEV1 ≥ 50% pred after BD) or (FEV1 < 80% predicted after BD and ≥ 9% reversibility)
* The patient is monitored by the AC service of the SHL.
* The GP of the patient is willing to participate in the trial.
* Written informed consent of participant

Exclusion Criteria:

* Patients treated primary by a pulmonologist
* Patients currently participating in another respiratory intervention study
* When the GP considers it detrimental to the patient to participate in the study
* Serious other non-pulmonary diseases (or disease-stages) that are presumed to lead to "lost to follow-up" because of the severity of the disease course (like diseases with low survival rate or mental deterioration)
* Serious other pulmonary diseases that effect bronchial symptoms and/or lung function, e.g. sarcoidosis, lung cancer, lung fibrosis
* Illiteracy

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-03; Primary Completion 2007-02 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Disease-specific health related quality of life assessed with the Chronic Respiratory Questionnaire (CRQ-SR) | At baseline, after one year follow-up, and after two years follow-up

SECONDARY OUTCOMES:
Number of exacerbations; generic HRQoL (SF12); lung function indices; level of respiratory symptoms (MRC); satisfaction with the health care received (EuroPep); direct and indirect medical costs. | Yearly: SF12, MRC, exacerbations; At baseline and end of the trial: EuroPEP, lung function indices; Continues by general practitioner registration: costs and exacerbations
Moreover special attention will be paid to process evaluation (e.g, compliance to recommendations by general practitioner and patients). | half-yearly for general practitioners and yearly for patients

CONTACTS AND LOCATIONS:
Overall Officials: Tjard Schermer, PhD, Study Director — Radboud University Nijmegen Medical Centre, department of general practice; Lisette van den Bemt, MSc, Principal Investigator — Radboud University Nijmegen Medical Centre, department of general practice; Chris van Weel, MD PhD professor, Study Chair — Radboud University Nijmegen Medical Centre, department of general practice
Locations (1):
- Regional Diagnostic Centre, Etten-Leur, The Netherlands (SHL), Etten-Leur, Netherlands

REFERENCES:
- [Derived] van den Bemt L, Schermer TR, Smeele IJ, Boonman-de Winter LJ, van Boxem T, Denis J, Grootens-Stekelenburg JG, Grol RP, van Weel C. An expert-supported monitoring system for patients with chronic obstructive pulmonary disease in general practice: results of a cluster randomised controlled trial. Med J Aust. 2009 Sep 7;191(5):249-54. PMID 19740044
- See also: Website Radboud University Nijmegen Medical Centre — http://www.umcn.nl